CLINICAL TRIAL: NCT02650063
Title: A Pharmacokinetic Study of DE-117 Ophthalmic Solution in Healthy Adult Male Subjects - Phase I Study -
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 01171502
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Male Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DE-117 ophthalmic solution (Experimental)
  Interventions: Drug: DE-117

INTERVENTIONS:
Drug: DE-117

SUMMARY:
The purposes of this study are to evaluate the safety and plasma pharmacokinetics of DE-117 ophthalmic solution (one drop once daily for 7 days) in healthy male adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adult volunteers

Exclusion Criteria:

* Subjects with any history of severe diseases that preclude participation in this study for safety reasons
* Subjects with any diseases that preclude participation in this study for safety reasons

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve (AUC) | 7 days
Maximum plasma concentration (Cmax) | 7 days
Time to maximum plasma concentration (Tmax) | 7 days
Elimination half-life (T1/2) | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CPC Clinical Trial Hospital, Medipolis Medical Research Institute, Kagoshima, Japan